CLINICAL TRIAL: NCT05382416
Title: Evaluation of the SHARE! Peer Toolkit Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: Emotional Health Association (Unknown); California Department of Health Services (Other)
Responsible Party: Principal Investigator, Louis D. Brown, Associate Professor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: HSC-SPH-22-0294
Record Dates: First submitted 2022-05-16; First posted 2022-05-19 (Actual); Last update posted 2024-04-11 (Actual); Status verified 2024-04

CONDITIONS: Mental Health
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: SHARE! will advertise the availability of their Peer Toolkit training via their website, email distribution list, and to individuals who previously expressed interest. Participants who enroll in the study will be clustered by worksite. The worksites will be randomized to receive the training either first in the Summer or after follow-up data collection in the Fall.
Who Masked: Outcomes Assessor
Masking Description: Data collection and analysis will occur without knowledge of participant intervention condition.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Peer Toolkit Training (Experimental): Participants assigned to this arm will attend online or in-person trainings on the SHARE! Peer Toolkit, which requires 60 hours of time to be completed over 10 weeks.
  Interventions: Behavioral: SHARE! Peer Toolkit Training
- Wait-list Control (No Intervention): The wait-list control will continue practice as usual and not receive peer toolkit training until after the follow-up data collection.

INTERVENTIONS:
Behavioral: SHARE! Peer Toolkit Training — The SHARE! Peer Toolkit training is designed to improve the performance of peer workers in their provision of peer support. The training covers each of the 12 tools in the Peer Toolkit, which are taught through brief presentations followed by group discussions and interactive exercises to help people competently use each of the tools. Training sessions are typically two hours each, three times per week for 10 weeks.
  Arms: Peer Toolkit Training

SUMMARY:
SHARE! the Self-Help and Recovery Exchange will engage peer workers in their Peer Toolkit training, which is designed to improve the performance of peer workers in their provision of peer support. The Peer Toolkit training currently has a waitlist of peer workers interested in taking the course for professional development purposes. These peer workers and their supervisors will be invited to complete a web-based survey at baseline and 4-month follow-up. Peer workers will be randomly assigned to enroll in the Peer Toolkit training immediately or after the follow-up survey. Analyses will compare participants who had the opportunity to complete the training to those still waiting to start the training. This study will inform the use of the Peer Toolkit as a training mechanism to build the capacity of peer workers in the mental health workforce.

DETAILED DESCRIPTION:
SHARE! the Self-Help and Recovery Exchange will engage peer workers in their Peer Toolkit training, which is designed to improve the performance of peer workers in their provision of peer support. The training covers each of the 12 tools in the Peer Toolkit, which are taught through brief presentations followed by group discussions and interactive exercises to help people competently use each of the tools. The training is offered both online and in-person, requires 60 hours of time, and is typically completed over the course of 4 months. Participation in the training is optional.

The Peer Toolkit training currently has a waitlist of peer workers interested in taking the course for professional development purposes. These peer workers and their supervisors will be invited to complete a web-based survey at baseline and 4-month follow-up. Peer workers will be randomly assigned to enroll in the Peer Toolkit training immediately or after the follow-up survey. Analyses will compare participants who had the opportunity to complete the training to those who are still waiting to start the training. This study will inform the use of the Peer Toolkit as a training mechanism to build the capacity of peer workers in the mental health workforce.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be employed as a peer worker or as the supervisor of a peer worker participating in the study.
* Participants must be willing to attend the SHARE! Peer Toolkit Training, which takes 60 hours to complete.

Exclusion Criteria:

* Peer workers who do not receive pay and volunteer for less than 15 hours per week

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 272 (Actual)
Dates: Start 2022-05-19 (Actual); Primary Completion 2023-04-01 (Actual); Study Completion 2023-04-01 (Actual)

PRIMARY OUTCOMES:
Peer support skills as assessed by interview questions | 4 months
  Assessed by a set of 6 interview questions that ask participants to describe what they would do in six peer support situations. Each question is rated from 1 to 9-total score is calculated as the average of the scores on all questions, and total score ranges from 1 to 9, with 1 indicating poor peer support skills and 9 indicating exceptional peer support skills.

SECONDARY OUTCOMES:
Perceived empathic and social self-efficacy as assessed by a questionnaire | 4 months
  Assessed by a set of 11 likert scale questions that ask participants to rate their ability to be empathic in responding to others' needs or feelings and managing interpersonal relationships. Each question is rated from 1 to 5-total score is calculated as the average of the scores on all questions, and total score ranges from 1 to 5, with 1 indicating not well at all and 5 indicating very well.
Empathic and social efficacy as assessed by a questionnaire | 4 months
  Assessed by a set of 11 likert scale questions that ask participants' supervisors to rate participants ability to be empathic in responding to others' needs or feelings and manage interpersonal relationships. Each question is rated from 1 to 5-total score is calculated as the average of the scores on all questions, and total score ranges from 1 to 5, with 1 indicating not well at all and 5 indicating very well.
Job satisfaction as assessed by a questionnaire | 4 months
  Assessed by a set of 5 likert scale questions that ask participants about their level of agreement with statements about their job satisfaction. Each question is rated from 1 to 5-total score is calculated as the average of the scores on all questions, and total score ranges from 1 to 5, with 1 indicating strong disagreement with positive statements about job satisfaction and 5 indicating strong agreement with positive statement about job satisfaction.
Work-related burnout as assessed by a questionnaire | 4 months
  Assessed by a set of 7 likert scale questions that ask the participant for the frequency of certain burnout-related experiences at their job. Each question is rated from 1 to 5-total score is calculated as the average of the scores on all questions, and total score ranges from 1 to 5, with 1 indicating Never/Almost Never having certain burnout-related experiences at their job and 5 indicating Always having certain burnout-related experiences at their job.
Perceived social support as assessed by a questionnaire | 4 months
  Assessed by a set of 12 likert scale questions that ask participants about their level of agreement with statements reflecting supportive relationships with family, friends, and a special person. Each question is rated from 1 to 7-total score is calculated as the average of the scores on all questions, and total score ranges from 1 to 7, with 1 indicating very strongly disagree with statements reflecting supportive relationships with family, friends, and a special person and 7 indicating very strongly agree with statements reflecting supportive relationships with family, friends, and a special person.
Social isolation as assessed by a questionnaire | 4 months
  Assessed by a set of 6 likert scale questions that ask participants about their frequency of feelings related to social isolation. Each question is rated from 1 to 5-total score is calculated as the average of the scores on all questions, and total score ranges from 1 to 5, with 1 indicating never having feelings related to social isolation and 5 always having feelings related to social isolation.
Recovery as assessed by a questionnaire | 4 months
  Assessed by a set of 21 likert scale questions that ask participants how they feel about themselves and their lives. Each question is rated from 1 to 5-total score is calculated as the average of the scores on all questions, and total score ranges from 1 to 5, with 1 indicating strongly disagree with positive statements about self and 5 indicating strongly agree with positive statements about self.
Psychological well-being as assessed by a questionnaire | 4 months
  Assessed by a set of 18 likert scale questions that ask participants about their level of agreement with statements reflecting psychological well-being. Each question is rated from 1 to 7-total score is calculated as the average of the scores on all questions, and total score ranges from 1 to 7, with 1 indicating strongly disagree with statements indicating psychological well-being and 7 indicating strongly agree with statements indicating psychological well-being.
Work contributions as assessed by a questionnaire | 4 months
  Assessed by a set of 12 likert scale questions that ask participants' supervisors to rate participants productivity and work quality. Each question is rated from 1 to 7-total score is calculated as the average of the scores on all questions, and total score ranges from 1 to 7, with 1 indicating strongly disagree with positive statements about work contributions and 7 indicating strongly agree with positive statements about work contributions.

CONTACTS AND LOCATIONS:
Overall Officials: Louis D Brown, PhD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- SHARE! the Self-Help and Recovery Exchange, Culver City, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Please contact the Principal Investigator for more information.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: De-identified data from published studies will be available after publication
Access Criteria: Please contact the Principal Investigator for more information.